CLINICAL TRIAL: NCT06775314
Title: The Effectiveness and Safety of Cleanser Containing Triethyl Citrate, Pyruvic Acid, Combination Cream Containing Triethyl Citrate, Ethyl Linoleate, GT Peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic Acid and Spot Cream Containing Triethyl Citrate, Ethyl Linoleate, GT Peptide-10, Honokiol As Adjuvant Therapy for Mild to Moderate Acne Vulgaris
Brief Title: The Effectiveness and Safety of Cleanser Containing Triethyl Citrate, Pyruvic Acid, Combination Cream Containing Triethyl Citrate, Ethyl Linoleate, GT Peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic Acid and Spot Cream Containing Triethyl Citrate, Ethyl Linoleate, GT Peptide-10, Honokiol
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Collaborators: Indonesian Society of Dermatology and Venereology (Unknown); College of Dermatologist and Venereologist (Unknown); Indonesia Medical Education and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette, Sp.DVE, Subsp. D.K.E, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AKNICARE
Record Dates: First submitted 2025-01-13; First posted 2025-01-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; Triethyl citrate; Pyruvic acid; Ethyl linoleate; GT peptide-10; Salicylic acid 0,5%; Zinc lactate; Hyaluronic acid; Honokiol
MeSH Terms: conditions — Acne Vulgaris | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): this arm will receive placebo cleanser, placebo combination cream, and placebo spot cream every morning and evening, and then placebo cleanser, placebo combination cream and adapalene 0,1% every night
  Interventions: Drug: Adapalene 0,1% cream; Drug: placebo cleanser; Drug: placebo cream combination; Drug: placebo spot cream
- Treatment (Active Comparator): this arm will receive cleanser, containing Triethyl citrate, Pyruvic acid, combination cream, containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic acid, and spot cream, containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol, every morning and evening, and then cleanser, containing Triethyl citrate, Pyruvic acid, combination cream, containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic acid, and adapalene 0,1% cream every night
  Interventions: Drug: Cleanser; Drug: Combination cream; Drug: spot cream; Drug: Adapalene 0,1% cream

INTERVENTIONS:
Drug: Cleanser — Cleanser consist of Triethyl citrate and Pyruvic acid, will be given to subjects to be applied every morning, evening and night in group 2
  Arms: Treatment
Drug: Combination cream — combination cream consist of Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic acid will be given to subjects to be applied every morning, evening and night in group 2
  Arms: Treatment
Drug: spot cream — spot cream consist of Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol, will be given to subjects to be applied every morning and evening in group 2
  Arms: Treatment
Drug: Adapalene 0,1% cream — adapalene 0.1% cream will be given to subjects to be applied every night in group 1 and 2
Drug: placebo cleanser — placebo cleanser will be given to subjects to be applied every morning, evening and night in group 1
  Arms: Placebo
Drug: placebo cream combination — placebo cream combination will be given to subjects to be applied every morning, evening and night in group 1
  Arms: Placebo
Drug: placebo spot cream — placebo spot cream will be given to subjects to be applied every morning and evening in group 1
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to learn the effectiveness and safety of Cleanser containing Triethyl citrate, Pyruvic acid, Combination cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic acid 0,5%, Zinc lactate, Hyaluronic acid and Spot cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol as Adjuvant Therapy for Mild to Moderate Acne Vulgaris. This research aims to answer the main questions, those are :

1. How is the effectiveness of Cleanser containing Triethyl citrate, Pyruvic acid, Combination cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic acid 0,5%, Zinc lactate, Hyaluronic acid and Spot cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol as Adjuvant Therapy for Mild to Moderate Acne Vulgaris?
2. How is the safety of Cleanser containing Triethyl citrate, Pyruvic acid, Combination cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic acid 0,5%, Zinc lactate, Hyaluronic acid and Spot cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol as Adjuvant Therapy for Mild to Moderate Acne Vulgaris?

Participants are males and females between 15-50 years old. Participants will be examined by dermatologist, and will be photographed in five different positions, and also evaluated by janus facial analysis system. The participants are asked to use Cleanser containing Triethyl citrate, Pyruvic acid, Combination cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic acid 0,5%, Zinc lactate, Hyaluronic acid and Spot cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol as Adjuvant Therapy. The participants will be evaluated in 28, 56 and 84 days after the treatment.

DETAILED DESCRIPTION:
This study is a clinical study with randomized controlled trial design to learn the effectiveness and safety of Cleanser containing Triethyl citrate, Pyruvic acid, Combination cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic acid 0,5%, Zinc lactate, Hyaluronic acid and Spot cream containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol as Adjuvant Therapy for Mild to Moderate Acne Vulgaris. This study will be conducted in three Dermatology and Venereology Education Centers in Indonesia located in Jakarta (Rumah Sakit Pusat Angkatan Darat Gatot Soebroto), Padang (Rumah Sakit Umum Pusat Dr. M. Djamil), Bali (Rumah Sakit Umum Pusat Prof. Dr. I.G.N.G Ngoerah). Group 1 will receive placebo cleanser, placebo combination cream, and placebo spot cream every morning and evening, and then placebo cleanser, placebo combination cream and adapalene 0,1% every night. Group 2 will receive cleanser, containing Triethyl citrate, Pyruvic acid, combination cream, containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic acid, and spot cream, containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Honokiol, every morning and evening, and then cleanser, containing Triethyl citrate, Pyruvic acid, combination cream, containing Triethyl citrate, Ethyl linoleate, GT peptide-10, Salicylic Acid 0,5%, Zinc Lactate, Hyaluronic acid, and adapalene 0,1% cream every night. All participant will be evaluated in day 28, 56, and 84. Therapy evaluation will be assessed by dermatologist based on the Global Acne Severity Scale (GEA Score), Indonesia Acne Expert Meeting (IAEM Score), Clinician Erythema Assessment (CEA), Total of Inflammation and Non-Inflammation lesions, Acne Sequelae, facial skin analysis with Janus Skin Facial Analysis, and evaluation of quality of life using Acne-Quality of Life (Acne-QoL).

ELIGIBILITY:
Inclusion Criteria:

* Female and male aged 15-50 years
* mild to moderate acne vulgaris according to IAEM (Indonesian Acne Expert Meeting) scale and GEA ( Global Acne Severity) scale
* The subject is willing to participate in the study until it is finished

Exclusion Criteria:

* History of allergy to dermocosmetic products
* Undergoing other acne therapy, medication, or invasive action in the last month
* Pregnant or breastfeeding subjects

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of acne severity | Re-evaluation on day 28, 56 and 84 of therapy
  Based on global acne severity scale (GEA score). On a scale of 0-5, 0 indicates no lesion, while 5 indicates very severy acne
Change of acne severity | Re-evaluation on day 28, 56 and 84 of therapy
  Based on Indonesia Acne Expert Meeting scale (IAEM scale). the scale consists of mild, moderate and severe.
total of inflammation lesion and non inflammation lesion | Re-evaluation on day 28, 56 and 84 of therapy
  The total lesion will be examined by dermatologist
acne sequelae | Re-evaluation on day 28, 56 and 84 of therapy
  The acne sequelae will be examined by dermatologist
Quality of life | Re-evaluation on day 28, 56 and 84 of therapy
  Based on acne quality of life (Acne-QoL). Total score of acne-QoL is 0-114, the higher score interprets better quality of life of acne vulgaris patient
Erythema severity | Re-evaluation on day 28, 56 and 84 of therapy
  based on clinician erythema assessment scale (CEA scale). on the scale of 0-4. 0 indicates no erythema, while 4 indicates severe erythema
Facial analysis | Re-evaluation on day 28, 56 and 84 of therapy
  The facial analysis will be done by using janus facial analysis system

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Pusat Angkatan Darat Gatot Soebroto, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided